CLINICAL TRIAL: NCT06941363
Title: Salvage Ultrahypofractionated Postoperative External Radiotherapy For Biochemical Recurrence
Acronym: SUPERB
Status: Recruiting | Type: Observational
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Principal Investigator, Stefano Arcangeli, Associate Professor, University of Milano Bicocca
Other Study IDs: SUPERB
Record Dates: First submitted 2025-04-15; First posted 2025-04-23 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer (Post Prostatectomy)
Keywords: biochemical recurrence; salvage RT; toxicity profile; oncological outcomes; linac-based SBRT
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1 fx SDRT
  Interventions: Radiation: SDRT

INTERVENTIONS:
Radiation: SDRT — Salvage Single Dose Radiation Therapy (SDRT) to the prostate bed up to 17 Gy

SUMMARY:
Recently, the Radiation Oncology Department at Fondazione IRCCS San Gerardo dei Tintori has been renovated and has been equipped with cutting edge technologies to treat prostate cancer. Specifically, the now available technology can track organ motion in real time, thus allowing improved precision in radiation delivery, with increased protection of the surrounding organs at risk. These facilities have already enabled the kickoff of two prospective observational trials, the ABRUPT and the POPART, which are currently ongoing in the treatment of intact prostate and the biochemical recurrence, respectively. Taken together, these observations provide the basis for the prospective clinical study herein proposed. Patients enrolled in the study will undergo salvage single stereotactic RT to the prostate bed by means of image guided volumetric intensity-modulated arc technique (IGRT-VMAT) and state-of-the-art treatment-planning and quality assurance procedures, with emphasis on normal tissue sparing and and pinpoint delivery accuracy via the use of devices that ensure stability and beam location reproducibility

DETAILED DESCRIPTION:
Patients enrolled in this observational prospective trial undergo image-guided (IGRT) with volumetric-modulated arc radiotherapy (VMAT) using the same equipment, techniques, and treatment-planning procedures as per clinical practice. Eligible patients are those with persistently detectable PSA post-operatively or those developing biochemical recurrence after prostatectomy with initially undetectable PSA, without evidence of macroscopic local relapse and/or regional and distant metastases at restaging.

This trial aims to assess the toxicity profile of salvage single-fraction stereotactic radiotherapy (RT) to the prostate bed delivered using an IGRT-VMAT technique. The study is conducted using a two-stage design consisting of an initial dose-finding phase followed by a dose-expansion phase.

Stage 1 - Dose escalation and interim safety analysis. In the first stage, a rolling six dose-escalation design is used to evaluate the safety of 15 Gy, 16 Gy, and 17 Gy, each delivered in a single fraction. Patients are enrolled in cohorts of 3 to 6 patients per dose level. In accordance with the rolling six design, no more than six patients may be concurrently enrolled at a given dose level and considered at risk for dose-limiting toxicity (DLT) during the 90-day evaluation period.

The objective of this stage is to identify the maximum tolerated dose (MTD), defined as the highest dose associated with ≤1 DLT among 6 evaluable patients, with DLT defined as any grade ≥3 toxicity occurring within 90 days from treatment.

An interim safety analysis is planned after approximately 18 patients (ideally 6 per dose level) have been treated and evaluated.

Stage 2 - Dose expansion. Following the interim analysis, the study proceeds with a dose-expansion phase, enrolling additional patients to reach a total sample size of 50 patients. If all three dose levels are deemed tolerable, they will all be carried forward into this expansion phase in a balanced manner.

The sample size of 50 patients was calculated to provide a statistical power of 91.1% for the GU endpoint and 92.9% for the GI endpoint, with a two-sided alpha level of 0.05. The overall statistical power to reject the null hypothesis across both endpoints is 84.6%.

The null hypothesis (H₀) is based on acute toxicity rates reported in the NRG-GU003 phase III randomized trial for the hypofractionated post-prostatectomy radiotherapy (HYPORT) arm, which reported ≥G2 toxicity rates of 31.0% for GU and 22.5% for GI toxicity. The alternative hypothesis (H₁) is derived from prior studies of stereotactic body radiotherapy (SBRT) in the salvage setting, including the POPART and SCIMITAR trials, assuming toxicity rates of 12% for GU and 6% for GI toxicity.

Primary and secondary endpoints will be evaluated across the entire expanded cohort.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of male sex ≥ 18 years of age.
* Subjects have freely signed the pertinent informed consent before the beginning of the study

  * Adenocarcinoma of the prostate treated with radical prostatectomy (any type of radical prostatectomy is permitted including retropubic, perineal, laparoscopic or robotically assisted; there is no time limit for the date of radical prostatectomy)
  * Detectable post-prostatectomy PSA of ≥ 0.1 - < 2.0 ng/mL either (1) persistently detectable post-operatively or (2) developing biochemical recurrence after prostatectomy (initially undetectable)
  * No evidence of N1 and/or M1 disease assessed by PSMA PET-CT within 90 days prior to registration
  * Negative Magnetic Resonance Imaging (MRI) of the pelvis in case of equivocal evidence of local relapse on PSMA PET-CT
  * Androgen deprivation therapy (ADT) allowed as per physician's discretion
  * ECOG performance status of 0-1
  * Ability to complete the questionnaires

Exclusion Criteria:

* N1 and or M1 patients
* Macroscopic local relapse at pelvic MRI.
* Prior radiation of any kind to the prostate gland or pelvis
* Prior brachytherapy
* History of inflammatory colitis or other active severe comorbidities
* Patients who are on immunosuppressant medication

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with biochemical relapse following radical prostatectomy
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-05-02 (Actual); Primary Completion 2033-05 (Estimated); Study Completion 2033-05 (Estimated)

PRIMARY OUTCOMES:
Number of participants with acute treatment-related adverse events as assessed by CTCAE v. 5.0 | 3 months
  To prospectively evaluate the cumulative incidence of acute (< 90 days from the end of treatment) genitourinary (GU) and gastrointestinal (GI) treatment-related toxicities and adverse events. Toxicity assessments are performed at baseline, end of treatment, and at 1, 2, and 3 months after radiotherapy.

SECONDARY OUTCOMES:
Number of participants with late treatment-related adverse events as assessed by CTCAE v.5.0 | 1, 2 and 5 years
  To prospectively evaluate the cumulative incidence of late (≥ 6 months) genitourinary (GU) and gastrointestinal (GI) treatment-related toxicities and adverse events.
QUALITY OF LIFE (QOL) assessed by Expanded Prostate Cancer Index Composite (EPIC-CP) Questionnaire. For each domain minimum symptom score (=0) means best QOL and maximum symptom score (=12) means worst QOL | 3 months, 1, 2 and 5 years
  To measure symptom scores for each QOL domain (urinary incontinence, urinary irritative/obstructive, bowel, sexual) after SDRT by EPIC-CP Questionnaire
Number of participants with urinary incontinence assessed by International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF), ranging from 0 (best) to 21 (worst) | 3 months, 1, 2 and 5 years
  To assess urinary continence after postoperative SDRT using ICIQ-SF
Number of participants with erectile dysfunction assessed by International Index of Erectile Function Questionnaire ranging from 5 (worst ) to 25 (best) | 3 months, 1, 2 and 5 years
  To assess erectile function after postoperative SDRT using IIEF 5
Number of participants with biochemical relapse assessed by PSA (cut off 0.20 ng/mL) | 2 and 5 years
  To assess biochemical outcome after postoperative SDRT using serum PSA levels

CONTACTS AND LOCATIONS:
Locations (1):
- Radiation Oncology, Fondazione IRCCS San Gerardo dei Tintori (University of Milan Bicocca), Monza, Italy, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ma TM, Ballas LK, Wilhalme H, Sachdeva A, Chong N, Sharma S, Yang T, Basehart V, Reiter RE, Saigal C, Chamie K, Litwin MS, Rettig MB, Nickols NG, Yoon SM, Smith L, Gao Y, Steinberg ML, Cao M, Kishan AU. Quality-of-Life Outcomes and Toxicity Profile Among Patients With Localized Prostate Cancer After Radical Prostatectomy Treated With Stereotactic Body Radiation: The SCIMITAR Multicenter Phase 2 Trial. Int J Radiat Oncol Biol Phys. 2023 Jan 1;115(1):142-152. doi: 10.1016/j.ijrobp.2022.08.041. Epub 2022 Aug 23. PMID 36007724
- [Background] Dess RT, Sun Y, Jackson WC, Jairath NK, Kishan AU, Wallington DG, Mahal BA, Stish BJ, Zumsteg ZS, Den RB, Hall WA, Gharzai LA, Jaworski EM, Reichert ZR, Morgan TM, Mehra R, Schaeffer EM, Sartor O, Nguyen PL, Lee WR, Rosenthal SA, Michalski JM, Schipper MJ, Dignam JJ, Pisansky TM, Zietman AL, Sandler HM, Efstathiou JA, Feng FY, Shipley WU, Spratt DE. Association of Presalvage Radiotherapy PSA Levels After Prostatectomy With Outcomes of Long-term Antiandrogen Therapy in Men With Prostate Cancer. JAMA Oncol. 2020 May 1;6(5):735-743. doi: 10.1001/jamaoncol.2020.0109. PMID 32215583
- [Background] Burdett S, Fisher D, Parker CC, et al. LBA64 duration of androgen suppression with post-operative radiotherapy (DADSPORT): a collaborative meta-analysis of aggregate data. Ann Oncol. 2022;33(7):S1428-S1429
- [Background] Ferrario F, Franzese C, Faccenda V, Vukcaj S, Belmonte M, Lucchini R, Baldaccini D, Badalamenti M, Andreoli S, Panizza D, Magli A, Scorsetti M, Arcangeli S. Toxicity profile and Patient-Reported outcomes following salvage Stereotactic Ablative Radiation Therapy to the prostate Bed: The POPART multicentric prospective study. Clin Transl Radiat Oncol. 2023 Nov 25;44:100704. doi: 10.1016/j.ctro.2023.100704. eCollection 2024 Jan. PMID 38111610
- [Background] Lucchini R, Franzese C, Vukcaj S, Purrello G, Panizza D, Faccenda V, Andreoli S, Poli GL, Baldaccini D, Lo Faro L, Tomatis S, Cazzaniga LF, Scorsetti M, Arcangeli S. Acute Toxicity and Quality of Life in a Post-Prostatectomy Ablative Radiation Therapy (POPART) Multicentric Trial. Curr Oncol. 2022 Nov 30;29(12):9349-9356. doi: 10.3390/curroncol29120733. PMID 36547147
- [Background] Buyyounouski MK, Pugh SL, Chen RC, Mann MJ, Kudchadker RJ, Konski AA, Mian OY, Michalski JM, Vigneault E, Valicenti RK, Barkati M, Lawton CAF, Potters L, Monitto DC, Kittel JA, Schroeder TM, Hannan R, Duncan CE, Rodgers JP, Feng F, Sandler HM. Noninferiority of Hypofractionated vs Conventional Postprostatectomy Radiotherapy for Genitourinary and Gastrointestinal Symptoms: The NRG-GU003 Phase 3 Randomized Clinical Trial. JAMA Oncol. 2024 May 1;10(5):584-591. doi: 10.1001/jamaoncol.2023.7291. Erratum In: JAMA Oncol. 2024 Jun 1;10(6):833. doi: 10.1001/jamaoncol.2024.1062. JAMA Oncol. 2025 Dec 1;11(12):1555. doi: 10.1001/jamaoncol.2025.4707. PMID 38483412